CLINICAL TRIAL: NCT03342391
Title: CEGIR 7808: Use of Unsedated Transnasal Esophagoscopy (TNE) to Monitor Dietary Management of Eosinophilic Esophagitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0237
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Phase (Other): Treatment Phase will evaluate the effectiveness of Transnasal Esophagoscopy (TNE) as an acceptable form of monitoring Eosinophilic Esophagitis
  Interventions: Other: Transnasal esophagoscopy

INTERVENTIONS:
Other: Transnasal esophagoscopy — single food antigen introduction OR removal of topical swallowed steroid therapy followed by surveillance utilizing TNE

SUMMARY:
The purpose of this study is to test the effectiveness of utilizing Transnasal Esophagoscopy as a means of monitoring Eosinophilic Esophagitis patients.

DETAILED DESCRIPTION:
A participant with an established diagnosis of EoE who is undergoing Standard of Care treatment with a four or less food elimination diet (not including or counting foods restricted at time of EoE diagnosis) OR is on topical swallowed steroid therapy with any number of foods eliminated from the diet, is in histological remission, and has been recommended as part of Standard of Care to start a single new food introduction OR remove the swallowed steroid treatment by the subject's clinical allergist or gastroenterologist will be enrolled in the study. 14-17 days after the introduction of the clinically recommended single food antigen, a TNE will be performed to assess the esophageal mucosa. TNE will be performed every 2 weeks for six weeks (3 total TNE) to evaluate recurrence time of mucosal eosinophilia (>15 eos/HPF), other histological changes, and patient tolerance to serial TNE. At week 6 a sedated esophagoscopy will be offered as an alternative choice to TNE if the participant chooses.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be able to understand and provide informed consent/assent
2. Males and females ages 5-22 years of age
3. History of an established diagnosis of EoE
4. Recent EGD or TNE (with in past 1 year) showing EoE remission (e.g. <15 x eosinophils/hpf) and currently without significant symptoms attributed to EoE.
5. On a four food or less elimination diet not including or counting foods restricted at time of EoE diagnosis OR on swallowed topical steroid therapy with any number of foods eliminated from the diet.
6. Female subjects of childbearing potential must have a negative pregnancy test upon study entry
7. Female subjects with reproductive potential, must agree to use FDA approved methods of birth control for the duration of the study
8. Children and families have desire to reintroduce potential food allergens and either the food antigen has been recommended with plans for its introduction as part of Standard of Care by the child's allergist and/or gastroenterologist OR the swallowed topical steroid therapy has been recommended to be discontinued by the child's allergist and/or gastroenterologist.
9. Children and families willing to undergo unsedated serial TNE

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol
2. Bleeding disorder
3. Unwilling to undergo unsedated TNE
4. Unwilling or unable to come to hospital at least 3 times over 6 weeks.
5. Currently treated with a swallowed corticosteroid which is not being discontinued.
6. Treated with oral corticosteroids within 8 weeks of the start of the study.
7. More than one change is being made to the EoE treatment regimen (e.g., more than a single food is being reintroduced during the study period; the swallowed topical steroid is being discontinued at the same time a food is being introduced).
8. EoE has been symptomatic with clinically significant symptoms attributable to EoE including dysphagia, abdominal pain or vomiting in the period since endoscopy
9. The finding of uncontrolled cough, significant rhinorrhea or rhinitis obstructing nasal passages, oxygen saturations <92% (high altitude normal saturation), temperature >38 degrees Celsius, significant gastrointestinal illness within 1 week of TNE, or provider determination of significant illness during pre-procedure history and physical on the day that the TNE is planned.
10. Pregnancy, breast feeding or plans to become pregnant
11. Unable to complete study procedures including endoscopy.
12. Allergy to any material or medicine used for procedures
13. Use of investigational drugs within 16 weeks of participation
14. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 5 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Histological Improvement | 6 weeks
  To prospectively and serially evaluate the recurrence of esophageal eosinophilia (>15 eosinophils per high power field) after a clinical single food antigen introduction OR removal of swallowed topical steroid therapy by the subject's clinical allergist or gastroenterologist in children with EoE using unsedated Transnasal Endoscopy/Esophagoscopy.

SECONDARY OUTCOMES:
Endoscopic Appearances/Histological Findings | 6 weeks
  1. To identify serially the clinical (endoscopic appearances) and other histological findings (lamina propria fibrosis, mast cells, lymphocytes) associated with dietary food introductions OR swallowed topical steroid therapy removal in children with EoE.
Sample Size | 6 weeks
  2. To determine and evaluate mucosal sample size obtained during TNE (2.0 mm or 1.2 mm forceps) compared to that obtained during those same subjects' previous traditional sedated endoscopy/esophagoscopy (2.8 mm forceps).
Decision to participate | 6 weeks
  3. To assess family factors determining decision to complete TNE study and subject's satisfaction with serial TNE using the previously reported TNE Qualitative Questionnaire, the General Anxiety Disorder (GAD)-7 Anxiety Instrument and a structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Friedlander, M.D., Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Denver, Colorado, United States

REFERENCES:
- See also: Related info — http://www.rarediseasesnetwork.org/cms/CEGIR